CLINICAL TRIAL: NCT06779097
Title: A Prospective, Single-arm, Multicenter, Phase IV Study to Evaluate the Efficacy and Safety of Vunakizumab in Adults With Moderate-to-severe Plaque Psoriasis Who Have Converted From Other Biologics
Brief Title: Phase IV Study: Vunakizumab Efficacy and Safety in Moderate-to-severe Plaque Psoriasis
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-DER-RWS-002
Record Dates: First submitted 2025-01-07; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vunakizumab (IL-17A inhibitor) (Experimental)
  Interventions: Drug: Vunakizumab (IL-17A inhibitor)

INTERVENTIONS:
Drug: Vunakizumab (IL-17A inhibitor) — Vunakizumab (IL-17A inhibitor)

SUMMARY:
This is a prospective, single-arm, multicenter, Phase IV study of 1564 patients with moderate-to-severe chronic plaque psoriasis to evaluate the efficacy and safety of Vunakizumab in patients with moderate-to-severe plaque psoriasis who have converted from other biologics. To explore the efficacy of difficult-to-treat area, patient satisfaction and patient-reported outcomes (PRO).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old at the time of signing the informed consent, regardless of gender;
2. Diagnosed with moderate to severe plaque psoriasis;
3. The subject voluntarily signs informed consent before the start of any procedures related to the study, can communicate with the researcher smoothly, understands and is willing to strictly comply with the requirements of this clinical study protocol to complete the study;
4. Patients who have been treated with biologics for ≥12 weeks prior to screening and are in line with the biologics conversion recommendations of the Chinese Guidelines for the Treatment of Psoriasis Biologics and Small Molecule Drugs (2024 edition), and who have been screened and evaluated by researchers as eligible for biologics therapy.

Exclusion Criteria:

1. Patients previously treated with IL-17A inhibitors (IL-17Ai) had primary failure;
2. Patients who had previously used IL-17A inhibitors (IL-17Ai) and experienced drug-related adverse events leading to drug withdrawal;
3. Patients with severe hypersensitivity to the active ingredient or any excipients of Vunakizumab;
4. Fertile women (defined as all women with physical conditions necessary for pregnancy) and men who are pregnant or unwilling or unable to use highly effective birth control during the study period and within 20 weeks after the last receipt of the study drug;
5. Patients with clinically important active diseases, such as active tuberculosis, active hepatitis, and active malignant tumors;
6. Any other circumstances that the investigator believes will prevent the subject from following and completing the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1564 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved at least a 90% improvement from baseline in PASI scores by week 12 (PASI 90). | Three months
Proportion of subjects achieving sPGA 0/1 response at week 12. | Three months

SECONDARY OUTCOMES:
Proportion of subjects with PASI 75, PASI 90, PASI 100, sPGA 0/1, and sPGA 0 at week 4, 12, and 52. | One month， Three months，Twelve months
The time when subjects reached PASI 75 and PASI 90 within 12 weeks | Three months
The time when subjects reached PASI 75, PASI 90, PASI 100 within 52 weeks. | Twelve months
Changes in PASI scores relative to baseline at each visit during 52 weeks. | Twelve months
Response rates of ACR (American College of Rheumatology) 20, ACR50 and ACR70 at week 4, 12, 24 and 52. | One month， Three months， Six months，Twelve months

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided